CLINICAL TRIAL: NCT05305794
Title: Effect of Weekly GLP1 Agonist Treatment in "Double Diabetes": a Randomized Open-label Study
Brief Title: Effect of Weekly GLP1 Agonist Treatment in "Double Diabetes"
Acronym: TOLEDDO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BOUILLET PHRCI 2020
Record Dates: First submitted 2022-03-09; First posted 2022-03-31 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Double Diabetes
MeSH Terms: interventions — Insulin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental)
  Interventions: Drug: Insulin + semaglutide treatment; Biological: Biological check-up
- Control (Active Comparator)
  Interventions: Drug: Usual insulin treatment; Biological: Biological check-up

INTERVENTIONS:
Drug: Insulin + semaglutide treatment — Usual insulin treatment + semaglutide (0.25 mg/week for 4 weeks, then 0.50 mg/week for 4 weeks, then 1 mg/week for 18 weeks, i.e. a total duration of 26 weeks). Upon introduction of semaglutide (ozempic) treatment, insulin doses will be reduced by 10% (basal insulin, basal rate and bolus)
  Arms: Semaglutide
Drug: Usual insulin treatment — Usual insulin treatment
  Arms: Control
Biological: Biological check-up — at D0, D90 and D180

SUMMARY:
Between 16% and 22% of type 1 diabetic patients present a clinical and biological profile of insulin resistance favored by a family history of type 2 diabetes or metabolic syndrome. They constitute a group of patients with "double diabetes" since they have both true type 1 diabetes and inherited insulin resistance, typical of type 2 diabetes.

For several years, GLP1 agonists have been successfully used in the treatment of type 2 diabetes, leading to very significant improvements in glycemic control and weight loss.

Because of the insulin-sensitizing power of GLP1 agonists, the investigators hypothesize that they could reduce insulin resistance in patients with "double diabetes" and thus improve their glycemic control.

The investigators propose to use in this study semaglutide, the most recent and most potent GLP1 agonist (superiority demonstrated compared to exenatide LP and dulaglutide) and administered as a weekly subcutaneous injection (in contrast to liraglutide administered daily).

ELIGIBILITY:
Inclusion Criteria:

* Person who has given written consent
* Patient over 18 years of age
* Patient with type 1 diabetes confirmed by a C-peptide below laboratory standards
* Age at diagnosis < 35 years
* Treated with optimized insulin therapy (multi-injections or pump) for at least 1 year, having received specific therapeutic education on insulin dose adaptation.
* BMI (weight/height2) ≥ 27 Kg/m².
* At least one of the following criteria:

  * Family history of type 2 diabetes (parents, grandparents, uncles, aunts, brothers and sisters)
  * Family history of obesity (BMI>30 Kg/m2) (parents, grandparents, uncles, aunts, siblings)
  * Triglycerides > 1.50g/l (1.7mmol/l)
  * HDL< 0.5 g/l (1.29 mmol/l) in women, HDL<0.4 g/l (1.03 mmol/l) in men
* HbA1c ≥ 7.5% and < 12% in the 3 months preceding inclusion
* Having continuous glucose monitoring by a CGM (Holter Glucose Monitoring) system: Guardian, Dexcom or Free Style Libre
* For women of childbearing age: using an effective method of contraception until 2 months after the end of treatment. Effective contraception includes: hormonal contraception, intrauterine device, bilateral tubal occlusion, vasectomy and sexual abstinence

Exclusion Criteria:

* person not affiliated to national health insurance
* Pregnant, parturient or breastfeeding woman
* HbA1c ≥12% in the 3 months preceding inclusion.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy, confirmed by a fundus examination performed in the 6 months preceding the selection
* Person under a measure of legal protection (curatorship, guardianship)
* Renal insufficiency (GFR<30 ml/mn)
* Hepatic insufficiency (INR> 1.5)
* BMI >40 kg/m².
* History of bariatric surgery
* History of pancreatitis
* Allergy to the active substance or to one of the excipients of OZEMPIC®.
* Patients treated with GLP1 agonists or oral antidiabetics in the month preceding month prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of time spent within glycemic target range (0.70-1.80 g/l) | Change from baseline at Day 180

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France